CLINICAL TRIAL: NCT04688619
Title: Adolescents as Change Agents in the Incorporation of a Parental Component for a School Based Prevention Program, to Promote Self-care Behaviors, Self Esteem, and Media Literacy
Brief Title: Adolescents as Change Agents in the Incorporation of a Parental Component for a School Based Prevention Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tel-Hai Academic College
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Primary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention Program "young In Favor of Myself", active parents (Experimental): The program "young In Favor of Myself" will be delivered to adolescence aged 10-12, over 3 months. The program contains nine weekly, 90-min sessions that focus on Media literacy, self-esteem, self-image and body image. The parents will also participate by receiving activities to do with their children, given to the adolescents during the scool program. All participants will complete a self-report questionnaire at baseline, after the program ends, and three months after the completion of the program.
  Interventions: Behavioral: Prevention Program "young In Favor of Myself", active parents
- Prevention Program "young In Favor of Myself", passive parents (Active Comparator): The program "young In Favor of Myself" will be delivered to adolescence aged 10-12, over 3 months. The program contains nine weekly, 90-min sessions that focus on Media literacy, self-esteem, self-image and body image. The parents won't participate in the program, they will get only a brochure about Media literacy, self-esteem, self-image and body image. All participants will complete a self-report questionnaire at baseline, after the program ends, and three months after the completion of the program.
  Interventions: Behavioral: Prevention Program "young In Favor of Myself", no parental involvement

INTERVENTIONS:
Behavioral: Prevention Program "young In Favor of Myself", active parents — Prevention program: "young In Favor of Myself", with parent participation
  Arms: Prevention Program "young In Favor of Myself", active parents
Behavioral: Prevention Program "young In Favor of Myself", no parental involvement — Prevention program: "young In Favor of Myself", without parent participation
  Arms: Prevention Program "young In Favor of Myself", passive parents

SUMMARY:
Cluster-Randomized Clinical trial, which includes the development and activation of an intervention program among young adolescents and their parents. Adolescents will be the "change agents" and will receive activities and assignments to complete together with their parents, as a mean for increasing parental involvement in the program. Study hypothesis is that the intervention program will yield improvement in adolescents whose parents participated in the program, in comparison with the adolescents whose parents weren't involved in the intervention. Results will be measured using the study questionnaire, to be filled out by the participants before, immediately after, and three months after the completion of the program. The questionnaire will include validated questionnaires with good psychometric qualities. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, received information about the program and the study and were asked to provide informed consent.

DETAILED DESCRIPTION:
Early adolescent (10-13 years) is characterized by hormonal changes and accelerated physiological growth. Significant risk factors for the physical and mental health of children and adolescents include, among other things, disordered eating patterns, overweight and reduced physical activity, low self-esteem and negative body image.

"In Favor of Myself" is a preventive intervention program. The program's primary goal is to increase adolescents' self-esteem and to prevent negative self-image and body image, as well as to development media literacy. In this study, the investigators will focus on the "Young In Favor of Myself " program, designed for ages 10-12, grades 5 and 6, and its main core is the development of self-care. To increase the effect of "Young In Favor of Myself " program on the adolescents, the investigators have developed a parental component in addition to the school-based activities. The adolescent participants will receive activities and assignments to complete together with their parents, making them the "change agents", with a goal of increasing parental involvement in the program. The study will first assess the parents' influence on the program, and then evaluate the difference in adolescent outcomes from the program with or without this supplement.

Results will be measured using the study questionnaire, to be filled out by the adolescent participants before, immediately after, and three months after the completion of the program. The questionnaire will include validated questionnaires with good psychometric qualities. Parents will complete a satisfaction questionnaire at the end of the program. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, received information about the program and the study and were asked to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of children 10-12 years old
2. 10-12-year-old children of participating parents
3. Participants who filled out the questionnaires before and after the program
4. Participants whose parents signed a letter of informed consent.

Exclusion Criteria:

1. Participants who didn't complete the questionnaires at baseline or at least twice.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Sociocultural Attitudes towards Appearance Questionnaire-4, Affects by Media subscale. | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  he Sociocultural Attitudes Towards Appearance Questionnaire (Schaefer et al., 2015). The investigators included the Media subscale, including 4 items. Items are rated on a 5-point scale: (1) always, (2) often, (3) sometimes, (4) rarely, (5) never. The total score is based on computing the average. A higher score indicates higher pressure from the media to change one's look.
Change from Baseline in Rosenberg Self Esteem Scale | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  Rosenberg Self Esteem Scale (Rosenberg, 1965)- 10 items. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or
  "strongly disagree" on items 1, 3, 4, 7, 10, and "strongly agree" or "agree" on items 2, 5, 6, 8, 9. Two or three out of three correct responses to items 3, 7, and 9 are scored as one item. One or two out of two correct responses for items 4 and 5 are considered as a single item; items 1,8, and 10 are scored as individual items; and combined correct responses (one or two out of two) to items 2 and 6 are considered to be a single item.
Change from Baseline in Body Esteem Scale | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  Body Esteem Scale- This questionnaire examines self-esteem of body and physical appearance and consists of 3 subscales: appearance (10 items), weight (8 items) and attribution 187 to others (5 items). Items are rated on a 5-point scale: (1) never, (2) rarely, (3) sometimes, (4) 188 often, and (5) always. A higher score indicates higher body-esteem (Mendelson, Mendelson, & White, 2001)
Change from Baseline in Eating Disorder Examination- Questionnaire (EDE-Q8) | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  Eating Disorder Examination- Questionnaire short version (EDE-Q8). The items are rated on a 6-point scale: (1) never, (2) rarely, (3) sometimes, (4) often, (5) usually, and (6) always. EDE-Q provides assessment of eating disorder psychopathology related to anorexia nervosa (AN), bulimia nervosa (BN), and binge-eating disorder (BED). (Kliem et al, 2016)
Change from Baseline in Advertising Scale | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  The Advertising scale contains 1 item- Identification of strategies used by media. This question is reflected as a protective factor. It contains 8 different strategies which participants choose from: higher number of strategies identified indicate better media literacy. (Golan et al., 2013).
Change from Baseline in Self-Caring | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  Developed by Prof. Moria Golan and assessed in previous research. Includes 14 items which are rated on a 4-point scale: (1) never, (2) rarely, (3) sometimes, (4) always. Items are summed, and higher scores indicate higher self-care behaviors. This questionnaire was designed to assess self care behaviors in adolescents.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic College of Tel Hai, Kiryat Shmona, North of Israel, Israel

IPD SHARING:
Plan to Share IPD: No